CLINICAL TRIAL: NCT06948513
Title: Effect of Over-the-counter Analgesics on Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zitelli & Brodland Skin Cancer Center (Other)
Responsible Party: Principal Investigator, Frank Lacy, Fellow, Zitelli & Brodland Skin Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1344913
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Naproxen; Acetaminophen; Standard of Care; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen (Experimental): These patients receive a one-time dose of naproxen at surgery completion. They are instructed to take acetaminophen as needed for additional pain
  Interventions: Drug: Naproxen; Drug: Acetaminophen (Standard of Care)
- Control (Active Comparator): These patients received 'standard of care' use of ibuprofen in combination with acetaminophen in a patient directed manner for pain control
  Interventions: Drug: Acetaminophen (Standard of Care); Drug: ibuprofen

INTERVENTIONS:
Drug: Naproxen — Naproxen given immediately post-operatively following Mohs surgery reconstruction
  Arms: Naproxen
Drug: Acetaminophen (Standard of Care) — Acetaminophen alternated with ibuprofen on an as needed, patient directed basis
Drug: ibuprofen — Ibuprofen alternated with acetaminophen in a patient directed manner for as needed pain control
  Arms: Control

SUMMARY:
In 2011, a randomized controlled trial compared acetaminophen, acetaminophen + ibuprofen, and acetaminophen + codeine for post-operative pain relief after Mohs surgery. In this study, the combination of acetaminophen + ibuprofen was shown to be superior to the other treatment groups at controlling postoperative pain. The study also detailed the timing at which patients experienced pain after cutaneous reconstruction, with peak pain scores occurring at 4 hours post-op for all three groups. Since its publication, the as needed dosage of acetaminophen alternated with ibuprofen has become the standard of care for most patients undergoing cutaneous reconstructive surgery. Additionally, studies from multiple disciplines including cutaneous surgery, emergency medicine, otolaryngology and obstetrics have found that use of non-steroidal anti-inflammatories pose no greater incidence of side effects.

Given that peak pain levels occur approximately four hours after cutaneous reconstruction, likely due to the cessation of lidocaine or other local numbing medications, patients may benefit from additional pain relief during this critical time period. However, it is standard practice to start acetaminophen and ibuprofen only as needed when pain begins. Further, given the short half-life of ibuprofen (2 hours), it is unlikely that this medication taken in the immediate postoperative period would be of benefit at the four hour time mark. Therefore, we theorize that the one-time dosage of a long-acting non-steroidal anti-inflammatory taken upon completion of cutaneous surgery may be superior to the as needed dosing of acetaminophen and ibuprofen.

DETAILED DESCRIPTION:
Upon completion of informed consent, enrolled participants will be randomized to one of two treatment groups.

Group 1 (intervention group): will receive a one-time, mandatory dose of Naproxen sodium 440 mg immediately following completion of cutaneous reconstruction. For a period of 24 hours after surgery, patients will then be instructed to use acetaminophen as needed per manufacturer instructions not to exceed 4 g in a 24 hour period. Patients will not be permitted to use additional nonsteroidal analgesics during the 24 hour period. Patients will be asked to record pain scales in a pain diary at time points 0, 2, 4, 6, 8, 10 and 24 hours after surgery as well as the amount and timing of breakthrough pain medication (acetaminophen). Patients will be contacted the day following their procedure by the Principal Investigator and their responses will be recorded. Upon recording of the patient's pain diary, their enrollment in the study is complete.

Group 2 (control group): will not receive any mandatory dose of postoperative analgesic. As is considered standard of care, these patients will be instructed to alternate use of ibuprofen and acetaminophen on an as needed basis per manufacturer instructions. The dose of acetaminophen is not to exceed 4 g in a 24 hour period. The dose of ibuprofen is not to exceed 1200 mg in a 24 hour period. Patients will be asked to record pain scales in a pain diary at time points 0, 2, 4, 6, 8, 10 and 24 hours after surgery as well as the amount and timing of breakthrough pain medication (acetaminophen or ibuprofen). Patients will be contacted the day following their procedure by the Principal Investigator and their responses will be recorded. Upon recording of the patient's pain diary, their enrollment in the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Mohs micrographic surgery with same-day reconstruction on the head/neck

Exclusion Criteria:

* Second intention wound healing Operative site not on head and neck Self-described allergies to acetaminophen or any non-steroidal anti-inflammatory medication Pre-existing pain condition requiring analgesics History of bleeding or clotting disorder Recent history of upper gastrointestinal bleeding or ulcers Advanced liver disease or renal impairment Pregnancy Current use of anticoagulant (examples: aspirin, clopidogrel, warfarin, apixaban)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patient reported pain score | 10 hours
  Recorded using a visual analog scale and taken at defined time intervals during postoperative period

SECONDARY OUTCOMES:
Additional pain medication used | 10 hours
  Amount of as-needed dosing taken by patients for pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Zitelli & Brodland Skin Cancer Center, Clairton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson H, Hildebolt C, Rowland K. Pain Relief with Combination Acetaminophen/Codeine or Ibuprofen following Third-Molar Extraction: A Systematic Review and Meta-Analysis. Pain Med. 2022 May 30;23(6):1176-1185. doi: 10.1093/pm/pnab334. PMID 34850186
- [Background] Sniezek PJ, Brodland DG, Zitelli JA. A randomized controlled trial comparing acetaminophen, acetaminophen and ibuprofen, and acetaminophen and codeine for postoperative pain relief after Mohs surgery and cutaneous reconstruction. Dermatol Surg. 2011 Jul;37(7):1007-13. doi: 10.1111/j.1524-4725.2011.02022.x. Epub 2011 May 11. PMID 21561527